CLINICAL TRIAL: NCT00147732
Title: A Multicentre, Randomised, Phase III Clinical Trial Comparing Accelerated Radiotherapy With Accelerated Radiotherapy Plus Carbogen and Nicotinamide (ARCON) in Clinical Stage T2-4 Laryngeal Carcinoma.
Brief Title: Randomized Trial of ARCON in Larynx Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 098; CKTO 2000-09
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Larynx Carcinoma
Keywords: larynx carcinoma; radiotherapy; carbogen; nicotinamide
MeSH Terms: conditions — Laryngeal Neoplasms

ARMS (2):
- 1 (Active Comparator): Accelerated radiotherapy
  Interventions: Radiation: Accelerated radiotherapy
- 2 (Experimental): ARCON
  Interventions: Radiation: ARCON

INTERVENTIONS:
Radiation: Accelerated radiotherapy — 68 Gy over 5.5 weeks
  Arms: 1
Radiation: ARCON — 68 Gy over 5.5 weeks Carbogen: 98% oxygen plus 2% carbon dioxide Nicotinamide 60 mg/kg daily
  Arms: 2

SUMMARY:
TITLE:

A multicentre, randomised, phase III clinical trial comparing accelerated radiotherapy with accelerated radiotherapy plus carbogen and nicotinamide (ARCON) in clinical stage T2-4 laryngeal carcinoma.

PRIMARY OBJECTIVE:

Does the addition of carbogen and nicotinamide to a schedule of accelerated radiotherapy in patients with clinical stage T2-4 laryngeal carcinoma improve local primary tumour control? Definitive analysis will be performed on local control rates at two years after completion of radiotherapy.

SECONDARY OBJECTIVES:

Does the addition of carbogen and nicotinamide

* increase the larynx preservation rate?
* increase the regional control rate?
* increase the toxicity of accelerated radiotherapy?
* improve the overall quality of life?
* improve the disease-free survival?
* improve the overall survival?

STUDY DESIGN:

An open-label, randomised clinical trial assigning patients in a 1:1 ratio to one of the following treatment arms:

* accelerated radiotherapy
* accelerated radiotherapy plus carbogen and nicotinamide

PATIENT CHARACTERISTICS AND NUMBER:

344 patients with clinical T2-4 laryngeal carcinoma

MEASUREMENTS:

* time to local failure
* time to regional failure
* survival with functional larynx
* overall and disease-free survival
* frequency and severity of complications related to radiotherapy and carbogen and nicotinamide
* quality of life assessment

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmed squamous cell carcinoma of the larynx.
* TNM-classification (UICC 1997, appendix I):
* T3-4 glottic or supraglottic carcinoma
* T2 glottic carcinoma with impaired cord mobility or subglottic extension
* T2 supraglottic carcinoma with invasion of mucosa of base of tongue or vallecula or invasion of the medial wall of the piriform sinus.
* any N-stage, M0.
* WHO performance status 0 or 1 (appendix II).
* Age > 18 years.
* Written informed consent.
* Quality of life questionnaire completed.

Exclusion Criteria:

* Prior or concurrent treatment for this tumour.
* Severe stridor and adequate debulking of airway not possible.
* Impaired renal function: serum creatinine above upper normal limit.
* Use of nefrotoxic medication (including ACE-inhibitors) that cannot be discontinued for the duration of the radiation treatment.
* Impaired hepatic function: ASAT and ALAT more than 1.5 times the upper normal limit.
* Use of anti-convulsants that cannot be discontinued for the duration of the radiation treatment.
* History of malignancy during the previous 5 years except basal cell carcinoma of skin, carcinoma in situ of the cervix, or superficial bladder neoplasm (pTa).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2001-04; Primary Completion 2008-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Local control | 2 years

SECONDARY OUTCOMES:
larynx preservation | 2 years
regional control rate | 2 years
toxicity | 5 years
quality of life | 2 years
disease-free survival | 5 years
improve the overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Johannes HA Kaanders, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (7):
- Netherlands (6):
  - Free University Medical Centre, Amsterdam
  - University Medical Centre Groningen, Groningen
  - Leids University Medical Centre, Leiden
  - Maastro Clinic, Maastricht
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - University Medical centre Utrecht, Utrecht
- Mount Vernon Hospital, Northwood, Middlesex, United Kingdom

REFERENCES:
- [Derived] Janssens GO, Langendijk JA, Terhaard CH, Doornaert PA, van den Ende P, de Jong MA, Takes RP, Span PN, Kaanders JH. Quality-of-life after radiotherapy for advanced laryngeal cancer: Results of a phase III trial of the Dutch Head and Neck Society. Radiother Oncol. 2016 May;119(2):213-20. doi: 10.1016/j.radonc.2016.02.023. Epub 2016 May 8. PMID 27165613
- [Derived] Janssens GO, Rademakers SE, Terhaard CH, Doornaert PA, Bijl HP, van den Ende P, Chin A, Takes RP, de Bree R, Hoogsteen IJ, Bussink J, Span PN, Kaanders JH. Improved recurrence-free survival with ARCON for anemic patients with laryngeal cancer. Clin Cancer Res. 2014 Mar 1;20(5):1345-54. doi: 10.1158/1078-0432.CCR-13-1730. Epub 2014 Jan 22. PMID 24452791